CLINICAL TRIAL: NCT06940921
Title: A Single-arm, Prospective Clinical Study of Low-dose Radiation Therapy (LDRT) Combined With Stereotactic Body Radiation Therapy (SBRT) and Cadonilimab for Advanced Gastric, Colorectal and Ovarian Cancers With Peritoneal Metastases
Brief Title: SBRT-LDRT-Cadonilimab for Advanced Gastric, Colorectal and Ovarian Cancers With Peritoneal Metastases
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhang Tao (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor-Investigator, Zhang Tao, Chief Physician, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhang Tao
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Advanced Gastric Cancer; Advanced Colorectal Cancer; Advanced Ovarian Cancer; Peritoneal Metastasis
Keywords: low-dose radiation therapy; stereotactic body radiation therapy; Cadonilimab; peritoneal metastasis; gastric cancer; colorectal cancer; ovarian cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Whole abdominal LDRT combined with SBRT followed by Cadonilimab group (Experimental): Patients in the experimental arm will receive stereotactic body radiation therapy (SBRT) to selected tumor sites and low-dose radiotherapy (LDRT) to the whole abdomen, followed by Cadonilimab immunotherapy.
  Interventions: Radiation: Low-Dose Radiation(LDRT) + Stereotactic body radiotherapy (SBRT); Drug: Cadonilimab

INTERVENTIONS:
Radiation: Low-Dose Radiation(LDRT) + Stereotactic body radiotherapy (SBRT) — Radiation: Stereotactic Body Radiation Therapy (SBRT)
  * Stereotactic Body Radiation Therapy (SBRT) will be performed first at a total dose of 20-50 Gy, delivered in 3-5 fractions of 6-10 Gy each. And the target area was specifically selected based on the location and size of the patient's tumor.
  Radiation: low-dose radiotherapy (LDRT)
  * Whole-abdominal low-dose radiotherapy will be initiated within 10 days of the end of SBRT with a total dose of 7-15 Gy at 0.5-2.0 Gy twice daily. And the target area included all suspicious tumor tissues and potential metastatic foci in the abdominal cavity.
Drug: Cadonilimab — · Cadonilimab: 6 mg/kg IV, D1, Q2W, until disease progression, death, toxicity intolerance or withdrawal of informed consent

SUMMARY:
The goal of this clinical trial is to see if high- and low-dose radiotherapy combined with immunotherapy can work in patients with advanced gastric, colorectal, and ovarian cancers with peritoneal metastases, and to learn about the safety of this new combination treatment modality. The main questions they aim to answer are:

* Can whole-abdominal low-dose radiotherapy (LDRT) combined with selected-site stereotactic body radiation therapy (SBRT) followed by Cadonilimab control peritoneal lesions and malignant ascites in patients with advanced solid tumors with peritoneal metastases?
* Can the novel treatment modality of high- and low-dose radiotherapy combined with immunotherapy produce a survival benefit in patients with advanced gastric, colorectal, and ovarian cancers who have received multiple lines of therapy?
* Is the safety profile of this new treatment modality acceptable?

Participants will:

* Receive stereotactic body radiation therapy (SBRT) to selected sites and low-dose radiotherapy (LDRT) to the whole abdomen, followed by bi-weekly treatment with Cadonilimab until disease progression, death, toxicity intolerance or withdrawal of informed consent.
* Receive whole body imaging and laboratory tests every 6-8 weeks to assess the efficacy of tumor treatment.

DETAILED DESCRIPTION:
Several studies have confirmed that the prognosis for advanced solid tumors for which there is no longer a standard of care is extremely poor, with optimal supportive care and an overall survival time of usually 1-5 months, and better treatment options are urgently needed to benefit patients' survival. For advanced solid tumors with peritoneal metastases, the prognosis is even worse. The peritoneal metastatic lesions respond poorly to chemotherapy, targeting, immunotherapy, surgical treatment, and other currently used treatments, and the expected survival time is short, so there is an urgent need to seek more effective treatment modalities.

There is a synergistic effect between radiotherapy and immunotherapy, and several studies have explored the combination of radiotherapy and immune checkpoint inhibitors in the treatment of solid tumors, and the results have shown that this combination regimen has a good anti-tumor effect, but the optimal radiotherapy modality and dose of radiotherapy are still in the exploratory stage. At present, some preclinical studies and small sample studies have shown that the combination of high- and low-dose radiotherapy can change the tumor immune microenvironment, reverse the state of immunosuppression, and play a strong anti-tumor effect in combination with immune checkpoint inhibitors.

Therefore, the investigators propose to conduct a single-arm, prospective clinical study of whole-abdominal low-dose radiotherapy (LDRT) combined with stereotactic body radiation therapy (SBRT) followed by Cadonilimab for the treatment of advanced gastric, colorectal, and ovarian cancers with peritoneal metastases. The study evaluates the efficacy of this combination therapy modality on peritoneal metastatic lesions, as well as the objective remission rate (ORR), disease control rate (DCR), duration of remission (DoR), progression-free survival (PFS), overall survival (OS), and safety of the patients. Our study aims to further explore the combination treatment options to improve the efficacy and prognosis of backline treatment for advanced tumors, and to provide more evidence for the clinical practice of radiotherapy combined with immunotherapy in advanced gastric, colorectal, and ovarian cancers with peritoneal metastases.

ELIGIBILITY:
Inclusion Criteria:

* With his/her own consent and signed Informed Consent Form (ICF), willingness and ability to comply with planned visits, study treatments, laboratory tests and other experimental procedures.
* At the time of signing the ICF, the subject must be ≥ 18 years of age with a life expectancy of ≥ 12 weeks.
* Gastric, colorectal, or ovarian cancer diagnosed by pathologic histology or cytology. And accompanied by peritoneal metastasis confirmed by pathohistology or cytology or imaging (CT/MRI/PET-CT).
* Advanced or metastatic gastric cancer, colorectal cancer, ovarian cancer (AJCC/UICC stage IV) confirmed by imaging of the chest, abdomen and pelvis (CT/MRI/PET-CT).
* Previously received multiple lines of systemic antitumor therapy, no longer available or refused standard treatment.
* At least 1 measurable lesion other than the lesion to be treated with SBRT according to RECIST 1.1 criteria. For lesions that have received prior radiotherapy, only a definite progression of that lesion is considered a measurable lesion.
* An Eastern Cooperative Oncology Group physical status score (ECOG) of 0-1.
* Appropriate organ function based on the following laboratory test values obtained during the Screening Period: white blood cell count ≥ 3 x 109/L, neutrophil count ≥ 1.5 x 109/L, platelet count 75 x 109/L; serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase or aspartate aminotransferase or ≤ 2.5 x UNL (hepatic metastasis) subjects should be ≤ 5 x ULN), serum creatinine ≤ 1.5 x UNL.
* Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days prior to study entry and be willing to use a medically approved, highly effective contraceptive such as an IUD, birth control pills, or condoms for the duration of the study and for 3 months after the last dose of study drug. For male subjects whose partner is a female of childbearing age, they should be surgically sterilized or agree to use an effective method of contraception for the duration of the study and for a period of 3 months after the final study drug administration.
* No concurrent participation in other clinical trials during the study period.

Exclusion Criteria:

* Previous or concurrent other active malignant tumors. Except for malignant tumors that have received curative treatment and have been free of disease for more than 5 years or carcinoma in situ that can be cured by adequate treatment.
* Current gastrointestinal diseases such as duodenal ulcer, ulcerative colitis, intestinal obstruction, or other conditions that may cause bleeding or perforation of the gastrointestinal tract as determined by the investigator.

Other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator.

* Thrombotic or embolic events, such as cerebrovascular accident, pulmonary embolism, deep vein thrombosis, have occurred within 12 months prior to enrollment.
* Myocardial infarction, severe/unstable angina pectoris, NYHA class 2 or higher cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, and symptomatic congestive heart failure.
* Systemic antibiotic use for ≥ 7 days within 4 weeks prior to enrollment in the study or unexplained fever > 38.5°C during screening/prior to first dose will be excluded. Fever due to oncologic causes may be enrolled at the discretion of the investigator.
* presence of any prior treatment-induced, unabated adverse events Common Terminology Criteria (NCI CTCAE Version 5.0) Grade 2 or greater toxicity, excluding anemia, alopecia, and skin pigmentation.
* history of idiopathic pulmonary fibrosis, opportunistic pneumonia, drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia, active tuberculosis on chest computed tomography scan at screening.
* Human Immunodeficiency Virus (HIV) infection or known Acquired Immune Deficiency Syndrome (AIDS), untreated active hepatitis (Hepatitis B, defined as HBV-DNA ≥ 500 IU/ml; and Hepatitis C, defined as HCV-RNA above the lower limit of detection of the analytical method) or combination of Hepatitis B and Hepatitis C co-infection.
* symptomatic, untreated, or active progressive central nervous system (CNS) metastases Patients with CNS lesions treated and asymptomatic are eligible for this study if they meet all of the following criteria: measurable lesions exist outside the CNS as defined by RECISTv1.1; the patient does not have a history of intracranial hemorrhage or intraspinal hemorrhage; and the patient has not received stereotactic radiotherapy within the last 7 days prior to the start of study treatment. days prior to the start of study treatment; patients have not received stereotactic radiotherapy within 14 days prior to the start of study treatment, whole-brain radiotherapy within 14 days prior to the start of study treatment, or neurosurgical resection within days prior to the start of study treatment; and patients do not need to be on continuous corticosteroid therapy for CNS disease.
* Presence of an active or previous autoimmune disease or immunodeficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis. Exceptions are: patients with a history of autoimmune hypothyroidism who are receiving thyroid replacement therapy are eligible; patients with type I diabetes mellitus who are receiving an insulin regimen and are in glycemic control are eligible; patients with eczema, psoriasis, chronic lichen simplex, or vitiligo with only cutaneous symptoms are eligible if all of the following criteria are met: the rash must cover < 10% of body surface area; good disease control at baseline and require only topical weak corticosteroid therapy; and no acute exacerbation of the underlying disease within the past 12 months.
* have used systemic immunosuppressive medications within 2 weeks prior to the start of study treatment or anticipate the need for systemic immunosuppressive medications during study treatment, with the following exceptions: patients receiving short-term, low-dose systemic immunosuppressive medications or patients receiving a one-time pulse of systemic immunosuppressive medications may be eligible to participate in this study after obtaining confirmation of their participation from the Medical Monitor; patients receiving salt corticosteroids, inhaled or low-dose corticosteroids for the treatment of chronic obstructive pulmonary disease (COPD) or asthma, or patients receiving low-dose corticosteroids for the treatment of upright hypotension or adrenal insufficiency are eligible to participate in this study.
* known or suspected history of allergy to any of the relevant drugs used in the study.
* Pregnant or lactating women.
* Women of childbearing age or men of childbearing potential who are not using or refuse to use an effective non-hormonal contraceptive.
* subjects with other serious physical or mental illnesses or abnormal laboratory tests that may increase the risk of participation in the study or interfere with the results of the study, as well as subjects who, in the opinion of the investigator, are unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Peritoneal response rate | within 3 years after primary treatment
  The Peritoneal Cancer Index (PCI) score is currently the most commonly used and validated tool for assessing the extent of peritoneal metastasis and prognosis. The method is to divide the abdominal cavity into 9 partitions, the small intestine into 4 partitions, a total of 13 partitions, and each partition is assigned a score of 0~3 according to the lesion size (LS) seen intraoperatively. That is, the LS score for each of the 13 divisions was determined by intraoperative or radiologic imaging, with a total score of 39 points. In this study, imaging evaluations were performed every 8 weeks to assess the efficacy of peritoneal tumor lesions by abdominal DWI + T2 MRI or abdominal CT enhancement. PCI scores ranged from 0~39, with higher scores implying more peritoneal metastatic lesions. The peritoneal response was evaluated as effective if the PCI score decreased compared with baseline, stable if the PCI score remained unchanged, and ineffective if the PCI score increased.

SECONDARY OUTCOMES:
Objective response rate (ORR) | within 3 years after primary treatment
  The proportion of all subjects treated in the study who had a best overall response (BOR) of complete remission (CR) or partial remission (PR) according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) .
Disease Control Rate (DCR) | within 3 years after primary treatment
  The proportion of all subjects receiving study treatment who have a best overall response (BOR) of complete remission (CR), partial remission (PR), or stable disease (SD) as assessed by RECIST version 1.1. If CR or PR is achieved, subjects must be confirmed no less than 4 weeks (28 days) after the initial evaluation.
Duration of Response (DoR) | within 3 years after primary treatment
  The time from the first recording of confirmed remission (CR or PR) to the time of the first recording of disease progression (according to RECIST version 1.1) or death due to any cause, whichever occurs first. For those subjects who are alive and without disease progression at the time of analysis data cut-off, censoring will be performed on the date of the final tumor determination. DoR will be evaluated only for subjects who achieved a confirmed remission CR or PR.
Progression-free survival (PFS) | within 3 years after primary treatment
  Defined as the subject from enrollment to the date of the first documented tumor progression or the date of death from any cause, whichever occurs first.
Overall Survival (OS) | within 3 years after primary treatment
  Overall Survival (OS) was defined as the time between the start of enrollment and the death of the subject due to all causes. The OS of subjects who were alive at the last follow-up visit was counted as data censored at the time of the last follow-up visit. The OS of subjects who were lost to follow-up was counted as data censored at the time of last confirmed survival prior to the loss of follow-up. OS for data censoring was defined as the time from randomization grouping to censoring.
Adverse events (AEs) | within 3 years after primary treatment
  The safety parameters in this study included clinical symptoms, vital signs, physical examination, and laboratory tests. Observed adverse events (AEs) were evaluated with reference to the National Cancer Institute (NCI) AE Common Terminology Criteria Version 5.0 (NCI CTCAE Version 5.0), including type, incidence, severity, time of onset and end, whether it was a serious adverse event, relevance to the study drug, and regression.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Tao, PhD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No